CLINICAL TRIAL: NCT00990782
Title: CEPELA I Trial: Capsule Endoscopy for Post-Ablation Esophageal Lesion Assessment
Brief Title: Capsule Endoscopy for Post-Ablation Esophageal Lesion Assessment
Acronym: CEPELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-634
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Esophageal Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): PillCam ESO Capsule Endoscope - all patients receive capsule endoscopy before and after RFA procedure.
  Interventions: Diagnostic Test: PillCam ESO Capsule Endoscope

INTERVENTIONS:
Diagnostic Test: PillCam ESO Capsule Endoscope — Utilization of the PillCam ESO capsule endoscope to evaluate the condition of a patient's esophagus before and after RFA therapy to treat atrial fibrillation.

SUMMARY:
This study utilizes a disposable capsule endoscope (Pillcam ESO) to assess the condition of a patient's esophagus before and after the RFA procedure, as the injury rate to the esophagus has not been established.

DETAILED DESCRIPTION:
Patients undergoing radiofrequency ablation (RFA) therapy for atrial fibrillation, can sometimes experience insult or injury to the esophagus, due to the proximity of the esophagus to the RFA treatment area. This study utilizes a disposable capsule endoscope (Pillcam ESO) to assess the condition of a patient's esophagus before and after the RFA procedure, as the injury rate to the esophagus has not been established.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with persistent atrial fibrillation selected for radiofrequency ablation
* Adults aged 18 years and older
* Patients able to give informed consent

Exclusion Criteria:

* Patients under the age of 18
* Patient unable to or unwilling to swallow the capsule endoscopes
* Patients with cardiac pacemakers, implanted cardiac defibrillators or other implanted electro-medical devices
* Pregnant or lactating females
* Subjects with history of abdominal, pelvic, or bowel surgery within the past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Dodig, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PillCam ESO Capsule Endoscope: All patients receive capsule endoscopy before and after RFA procedure.
  PillCam ESO Capsule Endoscope: Utilization of the PillCam ESO capsule endoscope to evaluate the condition of a patient's esophagus before and after RFA therapy to treat atrial fibrillation.
Period: Overall Study
Arm/Group | PillCam ESO Capsule Endoscope
Started | 93
Completed | 88
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | PillCam ESO Capsule Endoscope
Number analyzed (Participants) | 88
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 65
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Esophageal Lesions Identified Using Capsule Endoscopy
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam ESO Capsule Endoscope
Number analyzed (Participants) | 88
Participants | 15

2. Secondary Outcome: Number of Participants With Capsule-identified Esophageal Injury Who Report Symptoms Post-RFA
Time Frame: 14 Days
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam ESO Capsule Endoscope
Number analyzed (Participants) | 15
Participants | 6

ADVERSE EVENTS:
Time Frame: 3 Months
Arm/Group | PillCam ESO Capsule Endoscope
All-Cause Mortality (participants affected / at risk) | 0/88
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 30/88
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PillCam ESO Capsule Endoscope (N=88)
Chest Discomfort (General disorders) | 20
Throat Pain (General disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Abdominal Pain (General disorders) | 1
Fever (General disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes